CLINICAL TRIAL: NCT04121000
Title: Effects of Patient Controlled Erector Spinae Block on Postoperative Pain in Video Assisted Thoracoscopic Surgery (VATS) : A Randomized Controlled Study
Brief Title: Patient Controlled Erector Spinae Block at VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, OZCAN PISKIN, MD, ASSOCIATED PROFESSOR, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-79-08/05
Record Dates: First submitted 2019-10-02; First posted 2019-10-09 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain
Keywords: Erector Spinae Block,; VATS
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The study will be a two-arm parallel assignment. One group will receive erector spinae block and the other will receive PCA.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Block for VATS Group (Experimental): 40 patients who had VATS will receive erector spinae block for postoperative pain management. All patients will receive IV Midazolam (0.05mg/kg) premediacation. Standard monitorization of EKG, non- invasive blood pressure and pulsoximeter will be done and recorded in every 5 minutes. After sedation and standard monitorization, 20 minutes before the induction and in the prone positon the ESB procedure will be done. 10 % povidon- iodin will be used for sterilization and the USG probe will be covered with sterile sheath. The block will be done at the 8th thoracic vertebra line. The USG probe will be replaced 2-3 cm lateral to the spinous process in sagittal plane. When the erector spinae muscle is identified in the USG the needle will be guided caudally.0.5-1 ml local anesthetics will be given in order to confirm the needle is in the right place. After confirmation with 20 mL %0.25 bupivacaine the procedure will be performed.
  Interventions: Procedure: VIDEO ASSISTED THOTACOSOPIC SURGERY
- Patient - Controlled Analgesia for VATS Group (Experimental): 40 patients who had VATS will receive IV PCA for postoperative analgesia managemnet.
  Interventions: Procedure: VIDEO ASSISTED THOTACOSOPIC SURGERY

INTERVENTIONS:
Procedure: VIDEO ASSISTED THOTACOSOPIC SURGERY — VATS

SUMMARY:
In this study our aim is to investigate the effects of continue erector spinae block on postoperative pain in patients who underwent thoracoscopic surgery.

DETAILED DESCRIPTION:
Open thoracic surgeries are very painful procedures. After these procedures multimodal analgesia methods such as NSAIDs, opioids, PCA (patient-controlled analgesia), infiltration analgesia and thoracal epidural block are frequently used. Of these methods thoracal epidural block is the gold standart, however this technique is very invasive and has a high risk for complications. Lately Video Assisted Thoracoscopic Surgery (VATS) has become more popular because it reduces the hospital stay and is less invasive, hence the thoracic epidural block for postoperative pain has become more questionable. In this study we aimed to investigate the effects of continue Erector Spinae Block (ESB) on postoperative pain after VATS. The study will include 80 patients.

40 patients will receive ultrasound (USG) guided ESB and 40 patients will receive PCA.

All patients will recive IV Midazolam (0.05mg/kg) premedication. Standard monitorization of EKG, non- invasive blood pressure and pulsoximeter will be done and recorded in every 5 minutes. Fentanyl (1-2 µg/kg), Propofol (2-3 mg/kg) and Rocuronyum (0,5-0,8 mg/kg) will be given in induction of general anesthesia. Volume -controlled ventilation will be secured to have the values O2 saturation >98% and en-tidal carbondioxide 30-35 mm-Hg. For the mainentanance of general anesthesia the minimal alveolar concentration of sevoflurane will be 1. After the surgery every patient will receive 1 gr paracetemol and 100 mg tramadol for postoperative pain. Furthermore every patient will receive 8 mg ondansetrone for postoperative nausesa.

After sedation and standard monitorization, 20 minutes before the induction and in the prone position the Erecor Spinae Block (ESB) procedure will be done. 10 % povidone - iodin will be used for sterilization and the USG probe will be covered with sterile sheath. The block will be done at the 8th thoracic vertebra line. The USG probe will be replaced 2-3 cm lateral to the spinous process in sagittal plane. When the erector spinae muscle is identifed in the USG the needle will be guided caudally. 0.5-1 ml local anesthetics will be given in order to confirm the needle is in the right place. After confirmation with 20 mL %0.25 bupivacaine the procedure will be performed. The patients' VAS scores will be evaluated at the 1st,3rd, 6th, 12th, and 24th hours and will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 20- 75
* ASA (American Society of Anesthesiologists) Score I-III
* Undergoing elective Video Assisted Thoracic Surgery

Exclusion Criteria:

* ASA Score IV and higher
* Patinets with neurological deficits
* Paitents who have major vascular damage at the same side
* Mentally retarded patients
* Patients with alcohol or drug addiction
* Patients who are allergic to local anesthetics
* Pregnancy
* Paitents with coagulopathy
* Patients with skin infection at the side of the procedure
* Patients with pneumothorax at the side of the procedure
* Patient with a pacemaker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Perioperative and postoperative analgesic needs of patients | Change in VAS scores at the first 48 hours
  Our primary outcome is to measure and identify the analgesic needs of the patients at the perioperative and postoperative period.In order to measure the analgesic needs Visual Analogue Scale will be used and patients' pain scores will be measured.

SECONDARY OUTCOMES:
side effect. | 1st, 4rd, 8th,12th, 24th, 36th and 48 th hours after the procedure.
  side effects of opioids

CONTACTS AND LOCATIONS:
Overall Officials: OZCAN PISKIN, Principal Investigator — Bulent Ecevit University
Locations (1):
- Zonguldak Bulent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No